CLINICAL TRIAL: NCT04751006
Title: Effects of Balance Exercise With or Without Gaze Stabilization Exercises on Clinical Outcomes in Elderly Patients With Chronic Dizziness:A Randomized Controlled Trial
Brief Title: Effects of Balance Training With Gaze Stabilization Exercises in Elderly Patients With Chronic Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-UOL-FAHS/718-XII/2020
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Chronic Dizziness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gaze Group (Experimental): Participants performed balance training with gaze stabilization exercises
  Interventions: Other: Gaze Stabilization Exercises
- Control Group (Other): Participants performed balance training with saccade eye exercises
  Interventions: Other: Balance Training

INTERVENTIONS:
Other: Gaze Stabilization Exercises — Gaze group performed balance exercises with gaze stability exercise.Gaze stability exercises included two types of exercises vestibular adaptation and substitution exercises. In Adaptation exercises individual need to fixate on a visual target during horizontal and vertical head movement with a purpose of increasing gaze stability and a long term gain to vestibular system. Subsitution exercises are planned to use other eye movement stratigies to substitute vestibular function and sustained visual fixation. During Substitution exercises individual need to perfomed eye head movement between target with a purpose of clear sighting during these tasks. Balance exercises consist of both static and dynamic balance exercises with weekly progression making balance exercises more challenging.
  Arms: Gaze Group
Other: Balance Training — Participants performed balance training with saccade eye exercises.balance exercises included both static and dynamic balance exercises with a purpose of increasing mobility and stability of a posture by weekly progression. These exercises included standing on firm and foam surface with eyes open or close, heel stand, toe stand, marching on firm surface, forward and backward walking with normal base of support with weekly progression. Each task was performed for 5 repetitions with weekly progression in each task.
  Arms: Control Group

SUMMARY:
Effects of balance training with and without gaze stabilization exercises on clinical outcomes in elderly patients with chronic dizziness: A Randomized Controlled Trial

DETAILED DESCRIPTION:
In older adults dizziness is a common condition which is associated with repeated falls, fear of falling, depression, anxiety and ultimately loss of independence during activities of daily living. The main objective of this research was to compare the effects of balance training with and without Gaze Stabilization exercises on clinical outcomes in elderly patient with chronic dizziness.Total 64 participants after referral from neurologist were recruited in this study. These participants were randomly assigned into two groups i.e. Group A (Gaze group) and Group B (control group) with 32 participants in each group by sealed envelope method. Gaze group performed balance exercises with gaze stability exercises. Gaze stability exercises are further classified as adaptation and substitution exercises. Adaptation exercises support long term changes with a purpose of decreasing symptoms and maintain postural stability. On the other hand the substitution exercises improving central preprogrammed movement of eyes. Basically gaze stability exercises are defined as habituation exercises which reduce the symptoms of provoking stimulus by continuous exposure to it whereas, group B performed balance exercises with saccade eye exercises.Balance training includes both static and dynamic balance exercises, aimed to improved balance and postural stability with gradually increasing to challenging task. Exercises in balance training included a) single leg balance on firm surface b) heel stand c) marching on firm surface d) toe stand e) tandem walk f) forward and backward walking from normal base of support to weekly progression and training from eyes open to eye close from stable to unstable surface. Berg Balance Scale, Disability Handicapped inventory and Activity Specific Balance Confidence Scale were used to measure outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric population
* Both Gender
* H/O chronic dizziness with normal vestibular function
* H/O age related balance impairment
* H/O impaired balance having a Berg Balance Scale (BBS) score between 35-45
* Participant have sufficient cognitive and communication skills

Exclusion Criteria:

* H/O insufficient communication skills to follow instructions
* H/O impaired vestibular function
* H/O Visual impairment
* H/O Severe hearing loss
* H/O mental disorder that could restrains the ability to concentrate during therapy
* H/O Other systematic diseases
* Any history of marked musculoskeletal impairment, lower limb injury, surgery other than age related changes and balance disorder due to other neurological conditions like Parkinsonism, stroke, multiple sclerosis etc. were excluded from the study

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 6 Weeks
  Balance was measured using Berg Balance Scale
Disability Handicapped Inventory | 6 Weeks
  Precieved Disability was measured using Disability Handicapped Invertory
Activity Specific Balance Confidence | 6 Weeks
  Risk of Fall Prevention was measured using Activity Specific Balance Confidence

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Nida Fatima, Principal Investigator — University of Lahore
Locations (1):
- Univeristy Of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Results of study

REFERENCES:
- [Background] Geraghty AWA, Essery R, Kirby S, Stuart B, Turner D, Little P, Bronstein A, Andersson G, Carlbring P, Yardley L. Internet-Based Vestibular Rehabilitation for Older Adults With Chronic Dizziness: A Randomized Controlled Trial in Primary Care. Ann Fam Med. 2017 May;15(3):209-216. doi: 10.1370/afm.2070. PMID 28483885
- [Background] Hall CD, Heusel-Gillig L, Tusa RJ, Herdman SJ. Efficacy of gaze stability exercises in older adults with dizziness. J Neurol Phys Ther. 2010 Jun;34(2):64-9. doi: 10.1097/NPT.0b013e3181dde6d8. PMID 20588090
- [Background] Jahn K. The Aging Vestibular System: Dizziness and Imbalance in the Elderly. Adv Otorhinolaryngol. 2019;82:143-149. doi: 10.1159/000490283. Epub 2019 Jan 15. PMID 30947233
- [Result] Maciaszek J, Osinski W. Effect of Tai Chi on body balance: randomized controlled trial in elderly men with dizziness. Am J Chin Med. 2012;40(2):245-53. doi: 10.1142/S0192415X1250019X. PMID 22419420